CLINICAL TRIAL: NCT06015152
Title: Comparison Of The Efficacy Of Tazarotene 0.045% Versus Halobetasol Propionate 0.01% Lotion For the Treatment of Scalp Psoriasis
Brief Title: Comparison Of Efficacy Of Tazarotene 0.045% Vs Halobetasol Propionate 0.01% Lotion For Treatment of Scalp Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Nazia Jabeen, Principal Investigator, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO.F.2-81/2022-GENL/251/JPMC
Record Dates: First submitted 2023-03-25; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Scalp Psoriasis
MeSH Terms: interventions — tazarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A Tazarotene 0.045% (Experimental): Topical tazarotene 0.045% and halobetasol Propionate 0.01% . TAZ is the first receptor-selective retinoid used externally to treat plaque psoriasis . The major metabolite of tazarotene, tazarotenic acid, is quickly formed after application and binds to retinoic acid receptors (RARs) in the nucleus. Tazarotenic acid has a weak affinity for retinoid X receptors and prefers to bind to RARs b and g.
  Halobetasol propionate is a medication used to treat scalp psoriasis. It is a form of topical corticosteroid, which means it works by suppressing the immune system and reducing inflammation.
  Interventions: Drug: Tazarotene 0.045% Topical Application Lotion [ARAZLO]
- GROUP B Halobetasol Propionate 0.01% (Experimental): Topical tazarotene 0.045% and halobetasol Propionate 0.01% . TAZ is the first receptor-selective retinoid used externally to treat plaque psoriasis . The major metabolite of tazarotene, tazarotenic acid, is quickly formed after application and binds to retinoic acid receptors (RARs) in the nucleus. Tazarotenic acid has a weak affinity for retinoid X receptors and prefers to bind to RARs b and g.
  Halobetasol propionate is a medication used to treat scalp psoriasis. It is a form of topical corticosteroid, which means it works by suppressing the immune system and reducing inflammation.
  .
  Interventions: Drug: Tazarotene 0.045% Topical Application Lotion [ARAZLO]

INTERVENTIONS:
Drug: Tazarotene 0.045% Topical Application Lotion [ARAZLO] — [ARAZLO]

SUMMARY:
Psoriasis is a serious, immune-driven illness that affects around 2% of the population and has a wide range of clinical manifestations 1-3 . Many patients have localized illness, and topical therapy can be an important part of treatment.

tazarotene is the first receptor-selective retinoid for the topical treatment of plaque psoriasis. On application, tazarotene is rapidly hydrolyzed to its main metabolite, tazarotenic acid, which binds to retinoic acid receptors (RARs) in the nucleus. Tazarotenic acid selectively binds to RARs b and g . The predominant type of RAR expressed in the human epidermis is RAR, indicating that it may be an important mediator of retinoid action in skin. .

DETAILED DESCRIPTION:
Topical Corticosteroids is commonly used in situations of mild to moderate disease severity. However, long-term safety is still an issue, especially when utilizing stronger formulations,which come with a higher risk of local cutaneous adverse events (AEs). Telangiectasia, suppression of the hypothalamic-pituitary-adrenal (HPA) axis, and skin shrinkage are some of these negative consequences. By regulating gene transcription, tazarotene normalizes abnormal keratinocyte differentiation, reduces epidermal hyperproliferation, and decreases inflammation, the three pathogenic factors in psoriasis, thereby producing a more normal expression of skin differentiation in psoriatic lesions

ELIGIBILITY:
Inclusion Criteria:

* Patients between 30-50 years of age, either gender presenting with scalp psoriasis as per operational definition will be included in the study.

Exclusion Criteria:

* pustular psoriasis or had used phototherapy, photochemotherapy, or systemic psoriasis therapy within the last four weeks (or biologics within the last three months).
* Used topical treatment within 14 days prior to the baseline visit or who were diagnosed with skin conditions that would interfere with the interpretation of results were also excluded.

pregnant women, women attempting to become pregnant, lactation

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
The efficacy of Tazarotene 0.045% in Scalp Psoriasis | Efficacy will be assessed after 02 weeks
  Efficacy will be assessed by using Investigator's Global Assessment score for scalp psoriasis which is typically a 5-point scale from 0 to 4, with 0 = Clear/No Disease, 1 = Almost Clear, 2 = Mild, 3 = Moderate and 4 = Severe.
  Mean diference of IGA score before and after treatment will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: PARISA SANAWAR, FCPS, Principal Investigator — JPMC; KHADIJA ASADULLAH, FCPS, Principal Investigator — JPMC; FAIZA INAM, FCPS, Principal Investigator — JPMC
Locations (1):
- JPMC, Karachi, Sindh, Pakistan